CLINICAL TRIAL: NCT06113575
Title: Practical Clinical Application of Accelerated Intermittent Theta Burst Stimulation for Major Depressive Disorder
Brief Title: Practical Application of Accelerated iTBS for MDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonder Behavioral Health and Wellness (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SW-001-22
Record Dates: First submitted 2023-10-27; First posted 2023-11-02 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Major Depressive Disorder; Major Depressive Disorder, Recurrent Episode, Severe; Major Depressive Disorder, Recurrent, Moderate
Keywords: rTMS; Depression; MDD; TMS; iTBS; Accelerated; Theta Burst
MeSH Terms: conditions — Depressive Disorder, Major; Recurrence; Lymphoma, Follicular; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Scheduled Treatment Arm (Experimental): 5 day treatment course, 36 total treatments and clinical assessments.
  Interventions: Device: NeuroStar TMS

INTERVENTIONS:
Device: NeuroStar TMS — NeuroStar TMS treatment - 90-120% of Observed MT, 3 pulses/burst, 5 bursts/sec, 2 sec stimulation, 20 msec interval, 20 trains, 600 total pulses/session for 36 treatments in 5 days. 6 treatments on day 1, 8 treatments on days 2, 3, and 4, 6 treatments on day 5.

SUMMARY:
The goal of this observational study is to evaluate the feasibility and efficacy of accelerated iTBS in adults diagnosed with Major Depressive Disorder. The main question it aims to answer is:

What is the efficacy and tolerability of an accelerated iTBS regimen without radiological imaging in adults who have been diagnosed with Major Depressive Disorder and experience treatment resistant symptoms?

Participants will complete 36 iTBS treatments in an accelerated schedule over five days. They will also complete several clinical assessments throughout their enrollment to evaluate their depressive symptoms and response to treatment.

DETAILED DESCRIPTION:
The primary objective of this study is to demonstrate the preliminary effectiveness, tolerability, and feasibility of an accelerated, intermittent theta burst stimulation (iTBS) protocol for adults diagnosed with Major Depressive Disorder who are currently experiencing a Major Depressive Episode that does not rely on radiological imaging for the individualized targeting of desired treatment location of the dorsolateral prefrontal cortex and that is limited to 36 total treatments.

The study will be performed at a single site, where MDD patients, if eligible, can be consented to participate. Prior to iTBS Stimulation the Motor Threshold (MT) will be established for each subject individually. Each subject will be evaluated for 5 days during their iTBS treatment protocol and at 4 weeks post-treatment. The total study duration is expected to be approximately 8 months depending upon enrollment rate. The study consists of 8 visits. Each subject will be treated with an accelerated iTBS regimen for 5 days. This consists of 6-8 daily treatments which begin at 60-minute intervals for a total of 36 total treatments.

Visit 1 for subject intake with study physician. Visit 2 will consist of the establishment of baseline ratings. During visits 3-7 subjects will receive study protocol iTBS treatments. Visit 8 will be at 4 weeks post-treatment and will consist of administration of assessments. Study visits on treatment days are estimated to take between 5-7 hours depending on the day.

The Beam F3 System will be used to target the desired F3 location of the International 10-20 System. These coordinates are used to triangulate the desired treatment site on each patient on the first day of treatment and are saved for further treatments.

A Neuronetics NeuroStar XPLOR System version 3.6 will be used to deliver iTBS therapy. This consisted of 20 cycles of 5 bursts of 3 pulses at 50 Hz every 200 msec delivered in 2 second trains with an 8 second interval. Treatment sessions will be delivered hourly. Six or Eight sessions will be applied per day (3,600/4,800 pulses/day) for 5 consecutive days (21,600 pulses in total). Stimulation will not exceed 120% rMT.

Evaluations will consist of the Patient Health Questionaire-9 (PHQ-9), Quick Inventory of Depressive Symptomology (QIDS) Montgomery-Åsberg Depression Rating Scale (MADRS), Hamilton Depressive Ratings Scale (HAM-D). The primary endpoint is Change in MADRS scores from baseline to 4 weeks post treatment. Secondary endpoints include changes in the scores of all evaluations from baseline throughout the study. Response and remission rates will be calculated using both the MADRS and HAM-D at both the end of treatment and 4 weeks post study.

Staff handling data are trained in secure handling of Protected Health Information. Multiple layers of physical access will be employed, including individually assigned access cards and locked filing cabinets. Electronic records may be captured on the Sonder Wellness HIPAA compliant EMR database, Sonder Wellness managed and compliant shared network drive with controlled access to research staff, and/or a Sonder Wellness approved and secured external drive. All study data will exclusively use a de-identified code. Participant identifiers and corresponding code will be limited to key documents and maintained separately from the study data. Data will be collected and stored at a single site. Paper data will be stored on-site and electronic data on Sonder Wellness servers. Only Sonder Wellness research staff will have access to identifiable information. Data will be de-identified for affiliate analysis or summary reporting. No specimens will be collected or transported.

A sample size of 20 total subjects was selected as sufficient to perform a preliminary assessment of the effect size. The sample size is not based on formal power requirements for a statistical hypothesis test but is based on a desire to obtain a reasonable initial data set for exploratory and planning purposes.

All statistical analyses will be performed using SAS® version 9.4 (or higher). The full analysis set (FAS) will include all subjects who receive at least thirty treatment sessions. The FAS will be used for analyses of all efficacy outcome measures. The Safety population will include all subjects who receive at least one treatment session. This population will be used for demographic & Baseline characteristics and Safety outcome measures.

For efficacy endpoints, the Tables, Listings and Figures analysis and reporting will be performed on FAS population. A subject level listing will also be provided for each of these efficacy outcome MADRS, HAM-D, QIDS-16 and PHQ-9 separately presenting total score and each subscale score by different visits.

The primary endpoint of change in MADRS total score from baseline to 4 weeks post treatment will be analyzed using paired t test or Wilcoxon signed rank test. Mean change with the associated standard error and 95% CIs for the change will be presented along with the p-value.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* 22- 70 years
* Able to provide informed consent
* Diagnosed with major depressive disorder (MDD) and currently experiencing a major depressive episode (MDE)
* Subject failed to respond to at least one prior antidepressant medication
* Subject consented to receive TMS therapy to treat MDD with his or her physician independent of potential participation in this clinical study

Exclusion Criteria:

* Subject satisfies any one or more of the contraindications for TMS therapy per current treatment guidelines as determined by the PI
* Female with known or suspected pregnancy or is currently breastfeeding
* Total MADRS score of <20 at the screening or baseline visit
* Current diagnosis of a Substance Use Disorder (Abuse or Dependence, as defined by DSM-V-TR), with the exception of nicotine dependence
* History of schizophrenia or schizoaffective disorders, or any history of psychotic symptoms in the current or previous depressive episodes
* Any disorder which at screening is clinically predominant to their MDD or has been predominant to their MDD at any time within six months prior to screening
* Has a clinically significant abnormality on the screening examination that might affect safety, study participation, or confound interpretation of study results
* Participation in any clinical trial with an investigational drug or device within the past month or concurrent to study participation
* Any current or past history of any physical condition which in the investigator's opinion might put the subject at risk or interfere with study results interpretation
* Current use of opiates
* History of epilepsy
* History of shrapnel or metal in the head or skull
* History of cardiac event(s)
* History of OCD
* History of autism spectrum disorder
* History of rTMS exposure within 6 months of initial study treatment

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-11-23 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale | Baseline to four weeks post-treatment
  Change in Montgomery-Asberg Depression Rating Scale (MADRS) score, Minimum value = 0, Maximum value = 60. Higher score indicates a worse outcome.

SECONDARY OUTCOMES:
Patient Health Questionnaire | Baseline to four weeks post-treatment
  Change in Patient Health Questionnaire (PHQ-9) score, Minimum value = 0, Maximum value = 27. Higher score indicates a worse outcome.
Hamilton Depression Rating Scale | Baseline to four weeks post-treatment
  Change in Hamilton Depression Rating Scale (HAM-D) score, minimum value = 0, maximum value = 22. Higher score indicates a worse outcome.
Quick Inventory of Depressive Symptomatology | Baseline to four weeks post-treatment
  Change in Quick Inventory of Depressive Symptomatology (QIDS) score, minimum value = 0, maximum value = 27. Higher score indicates a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: John G. Luehr, MD, Principal Investigator — Sonder Behavioral Health and Wellness
Locations (1):
- Sonder Behavioral Health and Wellness, Minnetonka, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No